# Statistical Analysis Plan

Clinical Trial Number: 43CHSA1803

| | | <b>Table of Contents</b> | |
|---|---|---|---|
| 1 | | y Information | |
| | | Background | |
| | 1.1.1 | | |
| | 1.1.2 | | |
| | | Study objectives | |
| | 1.3 | Effectiveness assessments | |
| | 1.3.1 | | |
| | 1.3.2 | | |
| | 1.3.3 | Global Aesthetic Improvement Scale (GAIS) | 5 |
| | 1.3.4 | Subject satisfaction questionnaire | 6 |
| | 1.4 | Effectiveness endpoints | 7 |
| | 1.4.1 | Primary effectiveness endpoint | 7 |
| | 1.4.2 | Secondary effectiveness endpoints | 7 |
| | 1.5 | Safety assessments | 7 |
| | 1.6 | Safety endpoints | 8 |
| 2 | | stical Methods | |
| | | General methods | |
| | | Analysis Populations | |
| | | Study subjects | |
| | 2.3.1 | 3 | |
| | 2.3.2 | | |
| | 2.3.3 | | |
| | | Medical and surgical history, concomitant medication/procedures | |
| | | Effectiveness analysis | |
| | 2.4.1 | | |
| | 2.4.2 | | |
| | 2.4.3 | | |
| | 2.4.4 | | |
| | 2.5 | Safety Analysis | 12 |
| | 2.5.1 | Extent of exposure | 12 |
| | 2.5.2 | Subjects Diary | 13 |
| | 2.5.3 | Adverse events | 13 |
| | 2.6 | Interim Analysis | 13 |

Doc id

Print date:

MA-40407

2023-11-27 15:03

| 3 Pla | nned Tables and Figures | 15 |
|-------|-------------------------------------------------|----|
| 2.8 | Changes in the Analysis Planned in the Protocol | 14 |
| 2.7 | Determination of Sample Size | 13 |



# 1 Study Information

# 1.1 Background

# 1.1.1 Study design

This is a randomized, multi-center, evaluator-blinded, no-treatment controlled study of Sculptra for correction of Midface Volume Deficit and/or Midface Contour Deficiency in subjects of Chinese origin, men or women aged 18 years or older.

For Group A, after screening, eligible subjects will be treated from day 1 and followed up for 24 months.

For Group B, the study includes two phases as follows:

Main study phase: It is randomized, evaluator-blinded and no-treatment controlled. After screening, all eligible subjects will be randomized either to the Treatment Group or the Control Group in a 2:1 ratio. All the subjects will be followed up for 12 months.

Extension study phase: After the main study phase, the Treatment Group and Group A will be followed up for additional 12 months.

Each Treating Investigator will enroll 1 or 2 subjects as Group A. Before start of enrolment into Group B, the injection technique will be evaluated by the Sponsor or designee of Sponsor and performed after the subjects in Group A for each investigator have received their first treatment and second treatment. If treatments are found to be correctly performed, no further training is needed, there are no outstanding questions regarding the injection technique and no other corrective actions are identified, the enrolment in Group B can start for that investigator.

Each subject assigned to Group A and Treatment Group will receive up to 4 injection sessions with  $5 (\pm 1)$  weeks intervals. Study treatments should be stopped if optimal midface augmentation has been obtained or a maximum of 4 injection sessions completed. Optimal midface augmentation is defined as the best possible aesthetic result that can be obtained for an individual study participant, as agreed upon by the treating investigator and subject.

Subjects assigned to the Control Group will not receive treatment during the study.

For more details regarding the study, and references, see the Clinical Study Protocol (MA-39381).

#### 1.1.2 Number of subjects and randomization

The study will be performed at approximately 8 sites in China and approximately 32 subjects in Group A and 189 subjects in group B will be enrolled. Approximately 189 subjects in group B will be randomized in a 2:1 ratio to treatment with Sculptra (Treatment Group) or to no treatment (Control Group). The randomization list will be stratified by site.

#### 1.2 Study objectives

- To evaluate the effectiveness of Sculptra in the treatment of Midface Volume Deficit and/or Midface Contour Deficiency.
- To evaluate the safety of Sculptra in the treatment of Midface Volume Deficit and/or Midface Contour Deficiency.



#### Effectiveness assessments

For all assessments regarding subjects in Group A and subjects in Treatment Group in Group B, baseline will be defined as the observation that is closest to but prior to study treatment on Day 1. Likewise, change from baseline will be calculated as the value at a given time point minus the baseline value. For the Control Group baseline is defined as the observation that is closest to but prior to randomization.

# Medicis Midface Volume Scale (MMVS)

MMVS is a four-point scale assesses the fullness of the midface from Fairly Full (1) to Substantial Loss of Fullness (4) as described below. The blinded evaluator will rate the subject's right and left midface for severity of volume deficiency using the MMVS at screening, baseline, 6, 9, 12, 18 and 24 months in Group A and Treatment Group, and at screening, baseline 6, 9 and 12 months in Control Group. The treating investigator will do the MMVS evaluation at all visits in each group. The blinded evaluator and treating investigator will conduct their MMVS assessments using a photographic scale.

Table 1. Medicis Midface Volume Scale

| MMVS | |
|---|---|
| 1 | Fairly full midface; cheek prominence projected beyond the infraorbital rim at 45-degree view. |
| 2 | Mild loss of fullness in midface area; flatness of midface; cheek prominence at or behind infraorbital rim. May have slight presence of tear trough but not extending past mideye. Can start to see minimum volume loss of anterior cheek. |
| 3 | Moderate loss of fullness with slight hollowing below malar prominence; presence of the nasojugal groove extending past mideye. |
| 4 | Substantial loss of fullness in the midface area, clearly apparent hollowing below malar prominence; evidenced by significant indentation in the midface area. |

#### 1.3.2 3D Digital Imaging Analysis

The measurement of volume change in the midface (right and left combined) from baseline will be calculated by 3D digital image analysis at 6, 9, 12, 18 and 24 months in Group A and Treatment Group, and at 6, 9 and 12 months in Control Group.

#### Global Aesthetic Improvement Scale (GAIS) 1.3.3

The 5-graded Global Aesthetic Improvement Scale (GAIS) will be used to assess the aesthetic improvement of the midface fullness of both sides of the live subject as compared to photographs taken before treatment. Each midface side will be rated separately. The treating investigator and the subject will, independently of each other, respond to the question: "How would you describe the aesthetic improvement of the midface fullness for each side today compared to the photos taken before treatment?" GAIS will be assessed by treating investigator and subjects at each follow up visit.

Doc id 43CHSA1803 Statistical Analysis Plan - Sculptra China 👶 GALDERMA MA-40407

Table 2. Global Aesthetic Improvement Scale

| Rating | Definition (for treating investigator) |
|---|---|
| Very much improved | Optimal cosmetic result for the implant in this subject. |
| Much improved | Marked improvement in appearance from the original condition, but not completely optimal for this subject. |
| Improved | Obvious improvement in appearance from the original condition. |
| No change | The appearance is essentially the same as original condition. |
| Worse | The appearance is worse than the original condition. |

# Subject satisfaction questionnaire

Subjects will be asked about their satisfaction with the treatment outcome using a questionnaire at 6, 9, 12, 18 and 24 months in Group A and Treatment Group.

- 1). Do you think your Cheek Volume Deficit and/or Contour Deficiency has been improved with the treatment? Yes/No
- 2). Do you think that the overall result of the treatment looks natural? Yes/No

| 3). | Wo | ould you say that the study treatment? |
|---|---|---|
| | | Surpass your expectations Meet your expectations Do not meet your expectations You did not have any specific expectations before the injections |
| 4). | Do | you think that the treatment brings you more? (tick all boxes that apply) |
| | | Youth Beauty Harmony Symmetrical appearance Pep/Liveliness/Freshened look Self esteem /confidence |
| 5). | Wo | ould you say that you feel more attractive? Yes/No |
| 6). | Но | w do you feel about yourself since the treatment was performed? |

- 5).
- 6)

| Much better |
|-------------------------------------|
| Somewhat better |
| The Same |
| Worse; if worse, please explain why |

- 7). Overall, how satisfied are you with the treatment result?
  - Very satisfied Satisfied

Very much better

| | | Title 42 CHS A 1902 Statistical Analysis Plan Soulntre Chine | Doc id |
|---|---|---|---|
| ı | ♣ GALDERMA | 43CHSA1803 Statistical Analysis Plan - Sculptra China | MA-40407 |

| | | Somewhat satisfied |
|---|---|---|
| | | Not satisfied |
| 8). | Did | you get any feedback about your look from your family, friends, colleagues? |
| | | Positive feedback |
| | | Negative feedback |

- 9). Would you recommend this treatment to friends? Yes/No
- 10). Would you like to receive the same treatment again? Yes (exactly the same)/No

# 1.4 Effectiveness endpoints

□ No feedback

# 1.4.1 Primary effectiveness endpoint

Percentage of responders, defined by at least 1 point improvement from baseline on the MMVS on both sides of the face concurrently, as measured by the blinded evaluator at 12 months in both Treatment Group and Control group.

### 1.4.2 Secondary effectiveness endpoints

- Percentage of responders, defined by at least 1 point improvement from baseline on the MMVS on both sides of the face concurrently, as measured by the blinded evaluator at 6, 9, 18 and 24 months in Treatment Group, and at 6 and 9 months in Control Group.
- Percentage of responders, defined by at least 1 point improvement from baseline on the MMVS on both sides of the face concurrently, as measured by the treating investigator at 6, 9, 12, 18 and 24 months in Treatment Group, and at 6, 9 and 12 months in Control Group.
- Volume change from baseline over time of the right and left midface areas combined, as measured by digital 3D photography at 6, 9, 12, 18 and 24 months in Treatment Group, and at 6, 9 and 12 months in Control Group.
- Percentage of responders, defined by having "Improved", "Much improved" or "Very much improved" according to the Global Aesthetic Improvement Scale (GAIS) on both sides of the face combined, as assessed by the subject and the treating investigator at 6, 9, 12, 18 and 24 months in Treatment Group, and at 6, 9 and 12 months in Control Group.
- Percentage of subjects in each response category of each question in the subject satisfaction questionnaire in Treatment Group at 6, 9, 12, 18 and 24 months.

Note: Time of the Follow up visits at 6, 9, 12, 18 and 24 months is calculated from baseline/randomization.

#### 1.5 Safety assessments

The methods for collecting safety data are described in Section 8 of the Clinical Study Protocol (MA-39381) and include assessments of anticipated injection related reactions as collected in Subject Diary, Adverse Events (AE) and Serious Adverse Events (SAE). Laboratory assessments will be performed at screening for all subjects. In Group A and Treatment Group, it will also be taken at 12 months visit or at early termination if termination occurs before 12 months visit.



A two-point scale ("Yes" or "No" response) will be used for the causality assessments of AE and SAE. The Treating Investigator should be asked to indicate a response to each of the following questions in the eCRF:

"Do you consider that there is a reasonable possibility that the event may have been caused by the study product?"

"Do you consider that there is a reasonable possibility that the event may have been caused by the study product injection procedure?"

If any of these questions is answered with a 'Yes', the AE will be considered related. These assessments will also be reviewed by the Sponsor. In the case of a disagreement, the AE will be classified as "Related".

#### 1.6 Safety endpoints

- Incidence, intensity, duration, and onset of adverse events (AEs) collected throughout the study.
- Incidence, intensity, and number of days of anticipated injection related reactions, collected using 4-week subject diaries after each treatment session for the Treatment Group.

GALDERMA

Title
43CHSA1803 Statistical Analysis Plan - Sculptra China

MA-40407

#### **2** Statistical Methods

#### 2.1 General methods

All summaries for Group A and B will be done separately. The analyses described in the following sections primarily concern Group B. However, Group A will be analyzed in the same way, except that no hypothesis testing will be performed for Group A (there is only one treatment group in Group A), and the analyses will be done based on observed cases (i.e. no imputation of missing values will be done).

All statistical analyses, including summary tables and data listings, will be performed using the SAS® system (version 9.4 or later).

In general, effectiveness, safety, demography, subject characteristics, and treatment related variables will be presented using descriptive statistics. Continuous data will be summarized using n (number of observations), mean, standard deviation, median, minimum and maximum value, while categorical data will be presented by frequency and percentage. Graphs may be used as appropriate.

All statistical testing will be two-sided and performed at a significance level of 5%. Confidence intervals will be 2-sided and constructed using 95% confidence level.

If any SAP changes are needed before database lock (DBL), the SAP will be amended. Changes after DBL will be documented in the Clinical Study Report (CSR). If additional supportive or exploratory analyses are requested after SAP approval, this will not require amendment of the SAP, but these additional analyses will be described in the CSR. Some of the analyses detailed here may be more explicit or in some aspects different from those stated in the protocol. In case of differences, this SAP supersedes the statistical sections in the protocol.

All study data from the CRFs as well as derived variables will be provided in subject data listings.

#### 2.2 Analysis Populations

The following populations will be defined:

Safety

- Includes all subjects in Group B who were treated with Sculptra or randomized to no-treatment group. Subjects are analyzed based on the as treated principle.
- Full Analysis Set (FAS)
- Includes all subjects in Group B who were treated with Sculptra or randomized to no-treatment group. Subjects are analyzed according to the randomisation assignment.
- Per Protocol (PP)
- Includes all subjects in FAS that comply to the protocol procedures with no deviations that can affect the evaluation of the primary variable.

The FAS population is the primary population for all effectiveness analyses. All safety analyses will be based on the Safety population.

For Group A, all analyses will be performed based on all subjects.



#### 2.3 Study subjects

#### Subject disposition 2.3.1

The number of subjects in each study population (i.e. FAS, PP, and Safety) will be summarized by site and in total.

The disposition of subjects (including reasons for screening failures and withdrawals) will be presented by treatment group and in total. Subject accountability will be presented by treatment and visit.

#### 2.3.2 Withdrawals and Protocol deviations

All withdrawn subjects will be listed individually, including at least subject number, date and reason for withdrawal, and last visit performed. Subjects with CSP deviations will be listed individually, including subject number and observed deviation. Depending on the seriousness of the deviation, Group B subjects might be excluded from the PP population, which shall be documented prior to database lock.

For this study, the protocol deviations that will exclude Group B subjects from PP are identified (but not limited to) in Table 3 below.

Table 3. Protocol deviations

| | | Deviation |
|---|---|---|
| GENERAL | | |
| | | Visit out-of-window |
| | * | Follow-up at Month 12 after baseline performed earlier than 2 weeks before or later than 4 weeks after the scheduled visit for the treatment and control group |
| EFFECTIVENI | ESS | |
| | | Primary effectiveness endpoint |
| | * | No baseline MMVS by blinded evaluator available |
| | * | MMVS by blinded evaluator missing at Month 12 after baseline |
| | | Treatment |
| | * | Treatment not performed according to randomization |
| OTHER | | |
| | | Inclusion/exclusion criteria |
| | ÷ | Violate any inclusion or exclusion criteria considered to have<br>substantial effect on the primary effectiveness endpoint |
| | Concomitant medication/procedures | |
| | * | Take any prohibited concomitant medication/procedures considered to have substantial effect on the primary effectiveness endpoint |

Deviations from the SAP will be documented in the CSR.

GALDERMA

Title
43CHSA1803 Statistical Analysis Plan - Sculptra China

MA-40407

### 2.3.3 Demographic characteristics

Subject demographic and baseline characteristics data will be summarized for the FAS population by treatment group and in total.

# 2.3.4 Medical and surgical history, concomitant medication/procedures

All summaries will be done by treatment group based on the FAS population. Concomitant medications will be coded using the World Health Organization (WHO) Drug Dictionary. Medical History will be coded according to MedDRA.

The number and percent of subjects reporting medical history, and the number of events will be summarized by system organ class (SOC), in total and for ongoing events.

The number and percentage of subjects reporting concomitant medications will be summarized by treatment. In addition, the number and percent of subjects reporting concomitant medication, and the number of drugs (total number and the number of ongoing drugs), will be summarized by reason. The same summary will be done for concomitant procedures/treatments. Also, the number and percent of subjects, and the number of drugs, will be summarized by ATC code. Concomitant medications that started due to an AE will be summarized separately.

### 2.4 Effectiveness analysis

#### 2.4.1 Datasets analyzed

All effectiveness variables will be analyzed using the FAS population. The primary analysis will be repeated using the PP population. If it is deemed necessary, other analyses will be repeated using the PP population.

#### 2.4.2 Handling of missing data

Different assumptions regarding the missing data will be used. For the primary effectiveness analysis, missing values in the FAS will be assumed to be missing due to lack of effect. Therefore missing data up to the Month 12 visit will be imputed using the baseline observation carried forward (BOCF) method. As an alternative approach, missing data will be assumed to be unrelated to treatment effect. To impute data under this assumption, missing data up to the Month 12 visit will be imputed using the hot deck method. Both of these alternatives will estimate the effectiveness of the treatment policy (irrespective of use of not allowed treatments, procedures, or medications) rather than the true, clinical treatment effect.

To obtain an estimate of the true, clinical treatment effect, the primary effectiveness analysis will be performed using the PP population.

All other endpoints will be analysed on available data (observed cases - OC), i.e. no imputations will be done.

#### **Use of Hot Deck**

Each missing value in MMVS at Month 12 visit (recipient) will be imputed with a non-missing (observed) value from a subject randomly selected from the same imputation class (donor). Imputation classes will be defined based on treatment group (Sculptra or Control group), baseline MMVS value (2, 3 or 4 as assessed by the blinded evaluator) and age group (<55 vs. ≥55). Alternative imputation classes may be used if deemed necessary.

GALDERMA

Title

43CHSA1803 Statistical Analysis Plan - Sculptra China

MA-40407

### 2.4.3 Primary effectiveness analysis

The percentage of responders (a responder will be defined as a subject with at least 1 point improvement from baseline MMVS on both sides of the face concurrently) will be calculated at 12 months after baseline both in Treatment Group (denoted as  $\pi_{12M \text{ } Sculptra}$ ) and Control Group (denoted as  $\pi_{12M \text{ } Control}$ ) based on the blinded evaluator's assessment.

The null hypothesis H<sub>0</sub>:  $\pi_{12M \text{ Sculptra}} = \pi_{12M \text{ Control}}$  will be tested against the alternative hypothesis H<sub>1</sub>:  $\pi_{12M \text{ Sculptra}} \neq \pi_{12M \text{ Control}}$  by using a Fisher's exact test at a significance level of 5%. In addition, for each group and also for the difference between the two groups the two-sided 95% confidence intervals around the estimates of the percentage of responders will also be calculated. The treatment will be deemed a success if the p-value for the treatment difference on the primary endpoint is less than 0.05 (i.e. the proportion of responders is statistically significantly larger in the Treatment Group compared to the Control Group).

Subgroup analyses by site will be performed for the primary analysis. The difference in responder rates along with the 95% confidence intervals will be presented for each each site. No formal statistical testing will be carried out for the subgroup analysis.

In addition, to obtain an estimate of the true clinical treatment effect, the primary analysis will be rerun using the PP analysis set.

# 2.4.4 Secondary effectiveness analysis

The percentage of responders based on the MMVS on both sides of the face concurrently will also be derived at all applicable follow-up visits for both the blinded evaluator's assessment and the treating investigator's assessment respectively. The response rates and their 95% confidence interval will be presented by visit and group.

Fisher's exact test will be used to compare the response rates in the Treatment group versus the Control group based on the blinded evaluator's assessment and the treating investigator's assessment respectively. In other words, the null hypothesis

 $H_0$ :  $\pi_{t.Sculptra} = \pi_{t.Control}$  will be tested against the alternative hypothesis

 $H_1$ :  $\pi_{t,Sculptra} \neq \pi_{t,Control}$  for each of the timepoints t = Month 6 and Month 9 for the blinded evaluator's assessment, and t = Month 6, Month 9 and Month 12 for the treating investigator's assessment.

The volume change in the midface area as compared with baseline (right and left sides combined) obtained by 3D imaging will be presented descriptively by treatment for all applicable follow-up visits.

GAIS (by treating investigator and subject) and satisfaction with the treatment outcome will be analyzed descriptively.

#### 2.5 Safety Analysis

For Group B all safety variables will be summarized descriptively based on the safety population. For Group A all safety variables will be summarized descriptively based on all subjects.

#### 2.5.1 Extent of exposure

Data of extent of exposure and treatment procedure will be summarized per treatment session and also in total. Other relevant injection parameters, such as injection depth, injection method will be presented in a similar way.

GALDERMA

Title
43CHSA1803 Statistical Analysis Plan - Sculptra China

MA-40407

# 2.5.2 Subjects Diary

Number and percentage of subjects reporting anticipated injection related reactions, as collected in diaries will be presented in total and by maximum intensity for each treatment session (only Sculptra treated subjects). Graphs will be generated to illustrate the incidence over time. Number of days with the event will be summarized using mean, SD, min, max and median.

#### 2.5.3 Adverse events

All AEs will be coded according to MedDRA.

A summary of all AEs, by Treatment Group, will be provided, which will include:

- Number of subjects with at least one AE and number of events (in total as well as serious AEs)
- Number of subjects with at least one related AE and number of events (in total as well as serious AEs)
- Number of subjects with at least one unrelated AE and number of events (in total as well as serious AEs)
- Number of subjects who did not have an AE.

Related AEs as well as number of subjects with related AEs will be summarised by SOC, PT and intensity. In addition, for related AEs the number of days to onset and the duration of event will be summarised by SOC and PT using mean, SD, min, max and median. Action taken for related AEs will also be summarized. Related AEs will be summarized per treatment session.

Serious AEs will be listed.

Late onset (>21 days) AEs will be listed.

Related AEs with late onset (>21 days after most recent treatment) will be listed, if any.

Non-related AEs will be summarised by SOC, PT, and intensity and by Treatment Group.

Time to onset of an AE will be derived as the start date minus the date of most recent treatment. For the Control group date of randomization will be used instead of most recent treatment. If the start date is missing, it will be assumed that the AE started on the day of most recent treatment. If the start month is available but not the day, it will be assumed that the AE started on the first day of the month.

Duration of an AE will be derived as the stop date minus the start date + 1. If the start date is missing, it will be assumed that the AE started on the day of most recent treatment or date of randomization for the Control group. If the start month is available but not the day, it will be assumed that the AE started on the first day of the month. If the stop month is available but not the day, it will be assumed that the AE stopped on the last day of the month. Completely missing stop dates will not be imputed and therefore no duration will be calculated in these cases. Instead, the number of AEs that were ongoing at the end of the study will be given.

#### 2.6 Interim Analysis

An interim analysis will be performed when the month 12 visit is completed for all the subjects (main study phase).

#### 2.7 Determination of Sample Size

There are no available clinical data for Sculptra studied under conditions similar to the current study. However, based on what is seen in clinical studies of injectable fillers in the facial areas, it is

43CHSA1803 Statistical Analysis Plan - Sculptra China GALDERMA

Doc id

Print date:

MA-40407

2023-11-27 15:03

reasonable to assume a response rate of at least 60% in the Sculptra Treatment Group at Month 12. For the no treatment Control Group, response rate of 25.8% has been observed in an ongoing clinical trial in China. Based on this, it was assumed that the response rate will be maximum 30% in the no-treatment Control Group at Month 12.

With a sample size of 100 subjects treated with Sculptra and 50 subjects in the no-treatment control group, Fisher's Exact test will have approximately 90% power to detect difference between the anticipated percentage of responders at a 5% significance level (two-sided). To account for 20% drop-outs, approximately 126 will be randomized to the Sculptra group and approximately 63 to the control group.

#### 2.8 Changes in the Analysis Planned in the Protocol

Doc id 43CHSA1803 Statistical Analysis Plan - Sculptra China 👶 GALDERMA **MA-40407** 

#### 3 **Planned Tables and Figures**

# Group B:

Table 3-1 Analysis populations, by site

| Cit. | Subject<br>Id | Safety | | FAS | | PP | |
|-----------|---------------|--------|---|-----|---|----|---|
| Site | | n | % | n | % | n | % |
| Site 1 | | | | | | | |
| Site 2 | | | | | | | |
| Total (N) | | | | | | | |

<sup>% = (</sup>n/N)\*100

Table 3-2 Group A, by site

| te | Subject | Group A | |
|-----------|---------|---------|---|
| | Id | n | % |
| Site 1 | | | |
| Site 2 | | | |
| Total (N) | | | |

<sup>% = (</sup>n/N)\*100

Doc id

**MA-40407** 

Table 3-3 - Subject disposition, Group B

| Number of subjects | | Sculptra | Control | Total |
|----------------------------|-------------------|----------|---------|-------|
| Screened | | - | - | |
| Screening failures | | - | - | |
| Randomized | | | | |
| Treated | | | - | |
| Completed primary endpoint | | | | |
| Completed | | | | |
| Withdrawn | | | | |
| Reason for withdrawal | Withdrawn consent | | | |
| | Lost to follow-up | | | |
| | Medical reason | | | |
| | Other | | | |

<sup>%</sup> screening failures is based on total number of screened subjects.

In all other cases: % is based on the number of randomized subjects in each treatment group

Table 3-4 - Subject disposition, Group A

| Number of subjects | | Group A |
|-----------------------|-------------------|---------|
| Treated | | |
| Completed | | |
| Withdrawn | | |
| Reason for withdrawal | Withdrawn consent | |
| | Lost to follow-up | |
| | Medical reason | |
| | Other | |

👶 GALDERMA

43CHSA1803 Statistical Analysis Plan - Sculptra China

Doc id

Print date:

**MA-40407** 

2023-11-27 15:03

Table 3-5 Subject accountability, Group B

| Number of | | Scul | ptra | | Control | | | |
|---|---|---|---|---|---|---|---|---|
| subjects | Expected | Performed | Missed | Withdrawn | Expected | Performed | Missed | Withdrawn |
| Baseline /<br>Treatment 1 | | | | | | | | |
| Treatment 2 (optional) | | | | | | | | |
| Treatment 3 (optional) | | | | | | | | |
| Treatment 4 (optional) | | | | | | | | |
| Week 5 after last treatment | | | | | | | | |
| Month 6 after baseline | | | | | | | | |
| Month 9 after baseline | | | | | | | | |
| Month 12 after baseline | | | | | | | | |
| Month 18 after baseline | | | | | | | | |
| Month 24 after baseline | | | | | | | | |

Note: The main study consists of visits up to 12 months

Table 3-6 Subject accountability, Group A

| Number of subjects | Expected | Performed | Missed | Withdrawn |
|-----------------------------|----------|-----------|--------|-----------|
| Baseline / Treatment 1 | | | | |
| Treatment 2 (optional) | | | | |
| Treatment 3 (optional) | | | | |
| Treatment 4 (optional) | | | | |
| Week 5 after last treatment | | | | |
| Month 6 after baseline | | | | |
| Month 9 after baseline | | | | |
| Month 12 after baseline | | | | |
| Month 18 after baseline | | | | |
| Month 24 after baseline | | | | |

| ♣ GALDERMA | 43CHSA1803 Statistical Analysis Plan - Sculptra China | Doc id |
|---|---|---|
| | - Schortion Statistical Pinarysis Flair - Sculpti a Clinia | MA-40407 |

#### Table 3-7 Withdrawals, Group B

| Subject<br>Number | Treatment/Control | Date of withdrawal | Reason for withdrawal | Last visit | Date of last<br>visit |
|---|---|---|---|---|---|

# Table 3-8 Withdrawals, Group A

| Subject<br>Number | Date of withdrawal | Reason for withdrawal | Last visit | Date of last<br>visit |
|---|---|---|---|---|

# Table 3-9 – Protocol deviations affecting Per Protocol population (PP)

| Protocol deviation | Subject Number(s) | Number of deviations |
|--------------------|-------------------|----------------------|

# Table 3-10 – Protocol deviations not affecting Per Protocol population (PP), Group B

| Protocol deviation | Number of subjects |
|--------------------|--------------------|

# Table 3-11 - Protocol deviations, Group A

| Protocol deviation | Number of subjects |
|--------------------|--------------------|

Title
43CHSA1803 Statistical Analysis Plan - Sculptra China Doc id ♣ GALDERMA **MA-40407** 

# Group B

**Table 3-12** Summary of demographics and baseline characteristics, FAS

| Chamatariation | | Parameter | Group B | | |
|---|---|---|---|---|---|
| Characteristics | | Parameter | Sculptra | Control | Total |
| Age (years) | | n | | | |
| | | Mean (SD) | | | |
| | | Median | | | |
| | | Range | | | |
| Gender | | | | | |
| | Female | n (%) | | | |
| | Male | n (%) | | | |
| | Total | N | | | |
| Ethnic origin | | | | | |
| | Han<br>Chinese | n (%) | | | |
| | Other <sup>1)</sup> | n (%) | | | |
| | Total | N | | | |
| Baseline BMI | | n | | | |
| | | Mean (SD) | | | |
| | | Median | | | |
| | | Range | | | |
| MMVS<br>Blinded | Right side | | | | |
| | Score 2 | n (%) | | | |
| | Score 3 | n (%) | | | |
| | Score 4 | n (%) | | | |
| | Total | N | | | |
| MMVS<br>Blinded | Left side | | | | |
| | Score 2 | n (%) | | | |
| | Score 3 | n (%) | | | |
| | Score 4 | n (%) | | | |
| | Total | N | | | |

43CHSA1803 Statistical Analysis Plan - Sculptra China

**MA-40407** 

Doc id

Table 3-13: Subjects reporting medical history/concurrent diseases and number of conditions by MedDRA System Organ Class (SOC), FAS

| Primary SOC | Sculptra N = XX | | | | | | Control<br>N = XX | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Total | | Whereof ongoing at study start | | | Total | | | Whereof ongoing at study start | | |
| | Sub | jects | Number of | Subjects | | Number | Subjects | | | | Subjects | |
| | n | % | conditions | n | % | of conditions | n | % | of<br>conditions | n | % | of<br>conditions |
| Vascular disorders | | | | | | | | | | | | |
| Total | | | | | | | | | | | | |

 $\frac{1}{\%} = (n/N)*100$ 

Note: A single subject may have reported medical history/concurrent diseases by more than one primary SOC category

Table 3-14: Prior use of facial fillers or implants, FAS

| | | | culptra<br>= XX | Control<br>N = XX | | |
|-------|----------|---|-----------------|-------------------|----|------------|
| | Subjects | | Number of | | ts | Number of |
| | n | % | procedures | n | % | procedures |
| Total | | | | | | |

 $\frac{1}{\%} = (n/N)*100$ 

Note: A single subject may have had several fillers or implants

Print date: 2023-11-27 15:03

GALDERMA 43CHSA1803 Statistical Analysis Plan - Sculptra China

**MA-40407** 

Doc id

Table 3-15: Prior use of other facial dermatological procedures, FAS

| | | | culptra<br>= XX | $ \begin{array}{l} \text{Control} \\ N = XX \end{array} $ | | |
|---|---|---|---|---|---|---|
| | Subjec | ets | Number of | Subjects | | Number of |
| | n % | | procedures | n | % | procedures |
| Total | | | | | | |

 $\frac{\%}{(n/N)*100}$ 

Note: A single subject may have had several facial dermatological procedures

Table 3-16: Subjects reporting concomitant medication, FAS

| | | | lptra<br>XX | | Control<br>N = XX | | | |
|---|---|---|---|---|---|---|---|---|
| | N | lo | Y | es | N | o | Yes | |
| | n % n % | | | | n | % | n | % |
| Ongoing at study start | | | | | | | | |
| Initiated during study | | | | | | | | |
| Total | | | | | | | | |

 $<sup>\</sup>frac{1}{\%} = (n/N)*100$ 

Note: A single subject might have had concomitant medication ongoing at study start and initiated during study

Table 3-17: Subjects reporting concomitant medication and number of medications by reason, FAS

| | | | Sculptra<br>N = XX | | Control<br>N = XX | | | |
|---|---|---|---|---|---|---|---|---|
| Reason for concomitant medication | Sub | jects | Number of | f medications | Sub | jects | Number of medications | |
| incurcation | n | % | Total | Ongoing at study end | n | % | Total | Ongoing at study end |
| Related Adverse<br>Event | | | | | | | | |
| Unrelated Adverse<br>Event | | | | | | | | |
| Medical History | | | | | | | | |
| Other | | | | | | | | |
| Total | | | | | | | | |

 $<sup>\</sup>frac{1}{\%} = (n/N)*100$ 

Note: A single subject might have reported concomitant medication for several reasons

Table 3-18: Subjects reporting concomitant medication and number of medications by ATC code, FAS

| ATC | | | | ulptra<br>= XX | Control $N = XX$ | | |
|---|---|---|---|---|---|---|---|
| code | ATC text | Subjects Number of | | Subjects | | Number of | |
| | | n | % | medications | n | % | medications |
| Total | | | | | | | |

 $\frac{1}{\%} = (n/N)*100$ 

Note: A single subject may have reported several types of concomitant medication

#### Concomitant procedures

In a similar way as for conmed

# **Efficacy**

Table 3-19: MMVS responder rate at Month 12 by treatment (both sides of the face combined), Blinded Evaluator

| Donulation | Visit | Trantment | Subjects | Resp | onders | 95% C | Confidence | p-value |
|---|---|---|---|---|---|---|---|---|
| Population | VISIL | Treatment | N | n | % | in | interval | |
| FAS <sup>1)</sup> | Month 12 | Sculptra | | | | | | |
| | | Control | | | | | | |
| | | Difference | | | | | | |
| PP <sup>2)</sup> | Month 12 | Sculptra | | | | | | |
| | | Control | | | | | | |
| | | Difference | | | | | | |
| FAS <sup>3)</sup> | Month 12 | Sculptra | | | | | | |
| | | Control | | | | | | |
| | | Difference | | DOGE | | | | |

- 1) Note: Missing values at Month 12 are imputed using the BOCF method.
- 2) No imputation is used for PP analysis. Only subjects with complete data are included.
- 3) Note: Missing values at Month 12 are imputed using the Hot deck imputation method.

Note: Responder is defined as a subject with an improvement of at least one grade on the MMVS from baseline

Note: Responder rate (%) = (n/N)\*100

Note: P-values for the difference in proportions are based on the Fisher's Exact test.

Note: 95% confidence intervals are two-sided and calculated using the exact interval. For the difference, asymptotic confidence limits are used.

Doc id 43CHSA1803 Statistical Analysis Plan - Sculptra China 🚣 GALDERMA MA-40407

Table 3-20: MMVS responder rate over time (both sides of the face combined), Blinded Evaluator, FAS, OC

| <b>17:</b> -:4 | Toostoost | Subjects | Resp | onders | 95% Con | fidence | 1 |
|---|---|---|---|---|---|---|---|
| Visit | Treatment | N | n | % | inter | val | p-value |
| Month 6 | nth 6 Sculptra | | | | | | |
| | Control | | | | | | |
| | Difference | | | | | | |
| Month 9 | Sculptra | | | | | | |
| | Control | | | | | | |
| | Difference | | | | | | |
| Month 12 | Sculptra | | | | | | |
| | Control | | | | | | |
| | Difference | | | | | | |
| Month 18 | Sculptra | | | | | | |
| Month 24 | Sculptra | | | | | | |

Note: Responder is defined as a subject with an improvement of at least one grade on the MMVS from baseline.

Note: Responder rate (%) = (n/N)\*100

Note: P-values for the difference in proportions are based on the Fisher's Exact test.

Note: 95% confidence intervals are two-sided and calculated using the exact interval. For the difference, asymptotic confidence limits are used.

Figure 3-1: MMVS responder rate over time (both sides of the face combined), Blinded Evaluator, FAS, OC

Table 3-21: MMVS over time, Blinded Evaluator, FAS, OC

| | | | MMVS | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit / Trea | ntment | Side | 1 –<br>Fairly full | | | 2 –<br>Mild loss | | 3 –<br>Moderate loss | | 4 –<br>stantial<br>oss | Total |
| | | | n | % | n | % | n | % | n | % | N |
| Baseline | Sculptra | Left | | | | | | | | | |
| | | Right | | | | | | | | | |
| | Control | Left | | | | | | | | | |
| | | Right | | | | | | | | | |
| Month 6 | Sculptra | Left | | | | | | | | | |
| | | Right | | | | | | | | | |
| | Control | Left | | | | | | | | | |
| | | Right | | | | | | | | | |
| Month 9 | Sculptra | Left | | | | | | | | | |
| | | Right | | | | | | | | | |
| | Control | Left | | | | | | | | | |
| | | Right | | | | | | | | | |
| Month 12 | Sculptra | Left | | | | | | | | | |
| | | Right | | | | | | | | | |
| | Control | Left | | | | | | | | | |
| | | Right | | | | | | | | | |
| Month 18 | Sculptra | Left | | | | | | | | | |
| | | Right | | | | | | | | | |
| Month 24 | Sculptra | Left | | | | | | | | | |
| | | Right | | | | | | | | | |

 $\frac{0}{0} = (n/N)*100$ 

Note: The main study consists of visits up to 12 months

Table 3-22: MMVS responder rate over time (both sides of the face combined), Treating Investigator, FAS, OC Same as for Blinded Evaluator

Figure 3-2: MMVS responder rate over time (both sides of the face combined), Blinded Evaluator, FAS, OC

Table 3-23: MMVS over time, Treating Investigator, FAS, OC

Same as for Blinded Evaluator

Table 3-24: Volume change (mL) over time (both sides of the face combined) as measured by digital 3D photography, FAS

| Visit / Treatment | | N | Mean | SD | Median | Minimum | Maximum |
|-------------------|----------|---|------|----|--------|---------|---------|
| Month 6 | Sculptra | | | | | | |
| | Control | | | | | | |
| Month 9 | Sculptra | | | | | | |
| | Control | | | | | | |
| Month 12 | Sculptra | | | | | | |
| | Control | | | | | | |
| Month 18 | Sculptra | | | | | | |
| Month 24 | Sculptra | | | | | | |

Note: The main study consists of visits up to 12 months

Table 3-25: GAIS responder rate over time, (both sides of the face combined), Treating Investigator, FAS, OC

| Visit | Treatment | Subjects | Respo | onders | 95% C | onfidence |
|----------|-------------|----------|-------|--------|----------|-----------|
| VISIT | it Heatment | | n % | | interval | |
| Month 6 | Sculptra | | | | | |
| | Control | | | | | |
| Month 9 | Sculptra | | | | | |
| | Control | | | | | |
| Month 12 | Sculptra | | | | | |
| | Control | | | | | |
| Month 18 | Sculptra | | | | | |
| Month 24 | Sculptra | | | | | |

Note: Subjects with a GAIS rating of 'Very much improved', 'Much improved', or 'Improved' are defined as responders.

Note: Responder rate (%) = (n/N)\*100

Note: 95% Confidence Intervals are two-sided confidence intervals calculated using the exact interval.

Figure 3-3: GAIS responder rate over time, (both sides of the face combined), Treating Investigator, FAS, OC

Doc id 43CHSA1803 Statistical Analysis Plan - Sculptra China ♣ GALDERMA **MA-40407** 

Table 3-26: GAIS over time, Treating Investigator, FAS, OC

| | | | GAIS | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit / | Side | Very<br>imp | much roved | | luch<br>roved | Imp | roved | No c | change | Wo | orse | Total |
| Treatment | | n | % | n | % | n | % | n | % | n | % | N |
| Month 6 | Left | | | | | | | | | | | |
| Sculptra | Right | | | | | | | | | | | |
| Control | Left | | | | | | | | | | | |
| | Right | | | | | | | | | | | |
| Month 9 | Left | | | | | | | | | | | |
| Sculptra | Right | | | | | | | | | | | |
| Control | Left | | | | | | | | | | | |
| | Right | | | | | | | | | | | |
| Month 12 | Left | | | | | | | | | | | |
| Sculptra | Right | | | | | | | | | | | |
| Control | Left | | | | | | | | | | | |
| | Right | | | | | | | | | | | |
| Month 18 | Left | | | | | | | | | | | |
| Sculptra | Right | | | | | | | | | | | |
| Month 24 | Left | | | | | | | | | | | |
| Sculptra | Right | | | | | | | | | | | |

 $\frac{1}{\%} = (n/N)*100$ 

Note: The main study consists of visits up to 12 months

Table 3-27: GAIS responder rate over time (both sides of the face combined), Subject assessment, FAS, OC Same as for Treating Investigator

Figure 3-4: GAIS responder rate over time, (both sides of the face combined), Subject assessment, FAS, OC

Table 3-28: GAIS over time, Subject assessment, FAS, OC

Same as for Treating Investigator

Print date:

2023-11-27 15:03

Table 3-29: Subject Satisfaction Questionnaire, Question 1), Subjects randomized to Sculptra, FAS, OC

| Do you think your Cheek V | | it and/or Con<br>he treatment | | ncy has been | improved |
|---|---|---|---|---|---|
| Vigit (after begaline) | Y | es | N | lo | Total |
| Visit (after baseline) n % n % | | | | | |
| Month 6 | | | | | |
| Month 9 | | | | | |
| Month 12 | | | | | |
| Month 18 | | | | | |
| Month 24 | | | | | |

 $\frac{1}{\%} = (n/N)*100$ 

Note: The main study consists of visits up to 12 months

Table 3-30: Subject Satisfaction Questionnaire, Question 2), Subjects randomized to Sculptra, FAS, OC

| Do you think that | Do you think that the overall result of the treatment looks natural? | | | | |
|---|---|---|---|---|---|
| Vigit (after begaline) | Y | res | N | No | Total |
| Visit (after baseline) | n | % | n | % | N |
| Month 6 | | | | | |
| Month 9 | | | | | |
| Month 12 | | | | | |
| Month 18 | | | | | |
| Month 24 | | | | | |

 $\frac{1}{\%} = (n/N)*100$ 

Note: The main study consists of visits up to 12 months

Table 3-31: Subject Satisfaction Questionnaire, Question 3), Subjects randomized to Sculptra, FAS, OC

| Would you say that the study treatment: | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Visit (after baseline) | Surpass your expectations | | Meet your expectations | | Do not meet your expectations | | You did not have<br>any specific<br>expectations<br>before the<br>injections | | Total |
| | n | % | n | % | n | % | n | % | N |
| Month 6 | | | | | | | | | |
| Month 9 | | | | | | | | | |
| Month 12 | | | | | | | | | |
| Month 18 | | | | | | | | | |
| Month 24 | | | | | | | | | |

 $\frac{1}{\%} = (n/N)*100$ 

MA-40407

Doc id

Note: The main study consists of visits up to 12 months

Table 3-32: Subject Satisfaction Questionnaire, Question 4), Subjects randomized to Sculptra, FAS, OC

| | Do you think that the treatment brings you more: | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit You (after | uth | Beauty | | Harmony | | Symmetrical appearance | | Pep/Liveliness<br>/ Freshened<br>look | | Self-esteem/<br>confidence | | |
| baseline) | n | % | n | % | n | % | n | % | n | % | n | % |
| Month 6 | | | | | | | | | | | | |
| Month 9 | | | | | | | | | | | | |
| Month 12 | | | | | | | | | | | | |
| Month 18 | | | | | | | | | | | | |
| Month 24 | | | | | | | | | | | | |

 $\frac{1}{\%}$  = (n/N)\*100 where N=number of filled in questionnaires

Note: All that applies are ticked

Note: The main study consists of visits up to 12 months

Table 3-33: Subject Satisfaction Questionnaire, Question 5), Subjects randomized to Sculptra, FAS, OC

| Would you say that you feel more attractive? | | | | | |
|---|---|---|---|---|---|
| Visit (after baseline) | Y | res | N | Total | |
| | n | % | n | % | N |
| Month 6 | | | | | |
| Month 9 | | | | | |
| Month 12 | | | | | |
| Month 18 | | | | | |
| Month 24 | | | | | |

 $\frac{1}{\%} = (n/N)*100$ 

Doc id

Print date:

**MA-40407** 

2023-11-27 15:03

Table 3-34: Subject Satisfaction Questionnaire, Question 6), Subjects randomized to Sculptra, FAS, OC

| How do you feel about yourself since the treatment was performed? | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit (after baseline) | Very much better | | Much better | | Somewhat better | | The same | | Worse | | Total |
| | n | % | n | % | n | % | n | % | n | % | N |
| Month 6 | | | | | | | | | | | |
| Month 9 | | | | | | | | | | | |
| Month 12 | | | | | | | | | | | |
| Month 18 | | | | | | | | | | | |
| Month 24 | | | | | | | | | | | |

 $\frac{1}{\%} = (n/N)*100$ 

Note: The main study consists of visits up to 12 months

Table 3-35: Subject Satisfaction Questionnaire, Question 7), Subjects randomized to Sculptra, FAS, OC

| | Overall, how satisfied are you with the treatment result? | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Visit (after baseline) | Very satisfied | | Sati | Satisfied | | Somewhat satisfied | | Not satisfied | |
| | n | % | n | % | n | % | n | % | N |
| Month 6 | | | | | | | | | |
| Month 9 | | | | | | | | | |
| Month 12 | | | | | | | | | |
| Month 18 | | | | | | | | | |
| Month 24 | | | | | | | | | |

 $\frac{1}{\%} = (n/N)*100$ 

Note: The main study consists of visits up to 12 months

Table 3-36: Subject Satisfaction Questionnaire, Question 8), Subjects randomized to Sculptra, FAS, OC

| Did you get any feedback about your look from your family, friends and colleagues? | | | | | | | |
|---|---|---|---|---|---|---|---|
| Visit (after baseline) | Positive feedback | | Negative | feedback | No feedback | | Total |
| , | n | % | n | % | n | % | N |
| Month 6 | | | | | | | |
| Month 9 | | | | | | | |
| Month 12 | | | | | | | |
| Month 18 | | | | | | | |
| Month 24 | | | | | | | |

 $\frac{1}{\%} = (n/N)*100$ 

Table 3-37: Subject Satisfaction Questionnaire, Question 9), Subjects randomized to Sculptra, FAS, OC

| Would you recommend this treatment to friends? | | | | | |
|---|---|---|---|---|---|
| Visit (after baseline) | Y | es | N | Total | |
| | n | % | n | % | N |
| Month 6 | | | | | |
| Month 9 | | | | | |
| Month 12 | | | | | |
| Month 18 | | | | | |
| Month 24 | | | | | |

 $<sup>\</sup>frac{1}{\%} = (n/N)*100$ 

Note: The main study consists of visits up to 12 months

Table 3-38: Subject Satisfaction Questionnaire, Question 10), Subjects randomized to Sculptra, FAS, OC

| Would you like to receive the same treatment again? | | | | | |
|---|---|---|---|---|---|
| Visit (after begaling) | Y | es | N | No | |
| Visit (after baseline) | n | % | n | % | N |
| Month 6 | | | | | |
| Month 9 | | | | | |
| Month 12 | | | | | |
| Month 18 | | | | | |
| Month 24 | | | | | |

 $<sup>\</sup>frac{1}{\%} = (n/N)*100$ 

Doc id

Print date:

**MA-40407** 

# Treatment procedure

Table 3-39: Volume injected (both cheeks combined), Subjects randomized to Sculptra, Safety population

| Volume injected (mL) | | | | | | |
|------------------------|---|------|----|--------|---------|---------|
| Visit | N | Mean | SD | Median | Minimum | Maximum |
| Baseline / Treatment 1 | | | | | | |
| Treatment 2 (optional) | | | | | | |
| Treatment 3 (optional) | | | | | | |
| Treatment 4 (optional) | | | | | | |
| Total exposure | | | | | | |

Table 3-40: Treatment procedure (both cheeks combined, all treatments combined), Subjects randomized to Sculptra, Safety population

| Characteristic | Answer | Statistic | Result |
|---|---|---|---|
| Was 1 ml of lidocaine added to the vial before treatment? | Yes | n (%) | |
| | No | n (%) | |
| Local anaesthesia used? | Yes | n (%) | |
| | No | n (%) | |
| If local anaesthesia used | Topical cream | n (%) | |
| | Local infiltration | n (%) | |
| Needle gauge | 25 G | n (%) | |
| | 26 G | n (%) | |
| Depth of injection | Deep dermis | n (%) | |
| | Subcutaneous layer | n (%) | |
| | Supraperiosteal layer | n (%) | |
| | Other | n (%) | |
| Primary injection method | Linear Retrograde | n (%) | |
| | Serial Puncture | n (%) | |
| | Fanning | n (%) | |
| | Other | n (%) | |
| Post-treatment care (ice and massage) according to study protocol? | Yes | n (%) | |
| | No | n (%) | |
| Any deviation from the treatment procedure as | Yes | n (%) | |

| | Title |
|---|-------|
| ^ | 43CH |

# 13CHSA1803 Statistical Analysis Plan - Sculptra China

Doc id

Print date:

**MA-40407** 

2023-11-27 15:03

| Characteristic | Answer | Statistic | Result |
|----------------------------------|--------|-----------|--------|
| described in the study protocol? | | | |
| | No | n (%) | |

List deviations:...

Table 3-41: Treatment procedure (both cheeks combined), Subjects randomized to Sculptra, Safety population

| Characteristic | Visit | Statistic | Answer | Result |
|---|---|---|---|---|
| Was 1 ml of lidocaine added to the vial before treatment? | Baseline / Treatment 1 | n (%) | Yes | |
| | | n (%) | No | |
| | Treatment 2 (optional) | n (%) | Yes | |
| | | n (%) | No | |
| | Treatment 3 (optional) | n (%) | Yes | |
| | | n (%) | No | |
| | Treatment 4 (optional) | n (%) | Yes | |
| | | n (%) | No | |
| Local anaesthesia used? | Baseline / Treatment 1 | n (%) | Yes | |
| | | n (%) | No | |
| | Treatment 2 (optional) | n (%) | Yes | |
| | | n (%) | No | |
| | Treatment 3 (optional) | n (%) | Yes | |
| | | n (%) | No | |
| | Treatment 4 (optional) | n (%) | Yes | |
| | | n (%) | No | |
| If local anaesthesia used | Baseline / Treatment 1 | n (%) | Topical cream | |
| | | n (%) | Local infiltration | |
| | Treatment 2 (optional) | n (%) | Topical cream | |
| | | n (%) | Local infiltration | |
| | Treatment 3 (optional) | n (%) | Topical cream | |
| | | n (%) | Local infiltration | |
| | Treatment 4 (optional) | n (%) | Topical cream | |
| | | n (%) | Local infiltration | |
| Needle gauge | Baseline / Treatment 1 | n (%) | 25 G | |
| | | n (%) | 26 G | |

🚣 GALDERMA

Title
43CHSA1803 Statistical Analysis Plan - Sculptra China

Doc id

MA-40407

| Characteristic | Visit | Statistic | Answer | Result |
|---|---|---|---|---|
| | Treatment 2 (optional) | n (%) | 25 G | |
| | | n (%) | 26 G | |
| | Treatment 3 (optional) | n (%) | 25 G | |
| | | n (%) | 26 G | |
| | Treatment 4 (optional) | n (%) | 25 G | |
| | | n (%) | 26 G | |
| Depth of injection | Baseline / Treatment 1 | n (%) | Deep dermis | |
| | | n (%) | Subcutaneous layer | |
| | | n (%) | Supraperiosteal layer | |
| | | n (%) | Other | |
| | Treatment 2 (optional) | n (%) | Deep dermis | |
| | | n (%) | Subcutaneous layer | |
| | | n (%) | Supraperiosteal layer | |
| | | n (%) | Other | |
| | Treatment 3 (optional) | n (%) | Deep dermis | |
| | | n (%) | Subcutaneous layer | |
| | | n (%) | Supraperiosteal layer | |
| | | n (%) | Other | |
| | Treatment 4 (optional) | n (%) | Deep dermis | |
| | | n (%) | Subcutaneous layer | |
| | | n (%) | Supraperiosteal layer | |
| | | n (%) | Other | |
| Primary injection method | Baseline / Treatment 1 | n (%) | Linear Retrograde | |
| | | n (%) | Serial Puncture | |
| | | n (%) | Fanning | |
| | | n (%) | Other | |
| | Treatment 2 (optional) | n (%) | Linear Retrograde | |
| | · - / | n (%) | Serial Puncture | |
| | | n (%) | Fanning | |
| | | n (%) | Other | |
| | Treatment 3 (optional) | n (%) | Linear Retrograde | |
| | | n (%) | Serial Puncture | |

🚣 GALDERMA

Title
43CHSA1803 Statistical Analysis Plan - Sculptra China

Doc id

MA-40407

| Characteristic | Visit | Statistic | Answer | Result |
|---|---|---|---|---|
| | | n (%) | Fanning | |
| | | n (%) | Other | |
| | Treatment 4 (optional) | n (%) | Linear Retrograde | |
| | | n (%) | Serial Puncture | |
| | | n (%) | Fanning | |
| | | n (%) | Other | |
| Post-treatment care (ice and massage) according to study protocol? | Baseline / Treatment 1 | n (%) | Yes | |
| <u> </u> | | n (%) | No | |
| | Treatment 2 (optional) | n (%) | Yes | |
| | | n (%) | No | |
| | Treatment 3 (optional) | n (%) | Yes | |
| | | n (%) | No | |
| | Treatment 4 (optional) | n (%) | Yes | |
| | | n (%) | No | |
| Any deviation from the treatment procedure as described in the study protocol? | Baseline / Treatment 1 | n (%) | Yes | |
| | | n (%) | No | |
| | Treatment 2 (optional) | n (%) | Yes | |
| | | n (%) | No | |
| | Treatment 3 (optional) | n (%) | Yes | |
| | | n (%) | No | |
| | Treatment 4 (optional) | n (%) | Yes | |
| | | n (%) | No | |

List deviations:...

Print date:

2023-11-27 15:03

# Safety

Table 3-42: Anticipated injection related reactions recorded in the subject diary after first treatment (both sides of the face combined), Safety population

| | Treatment with Sculptra N=XX | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Event | C1- | : | | | Maximum | intensity | | |
| | Sub | jects | Mil | ld | Mod | erate | Sev | ere |
| | n | % | n | % | n | % | n | % |
| Pain | | | | | | | | |
| Tenderness | | | | | | | | |
| Localized redness | | | | | | | | |
| Bruising | | | | | | | | |
| Hematoma | | | | | | | | |
| Edema | | | | | | | | |
| Other | | | | | | | | |
| No diary<br>events | | | | | | | | |

% = (n/N)\*100

Note: Percentages for intensity categories are based on the number of subjects reporting the symptom.

Table 3-43: Number of days anticipated injection related reactions recorded in subject diary after first treatment (both sides of the face combined), Safety population

| Event | Treatment with Sculptra N=XX | | | | | |
|---|---|---|---|---|---|---|
| | n | Mean | SD | Minimum | Median | Maximum |
| Pain | | | | | | |
| Tenderness | | | | | | |
| Localized redness | | | | | | |
| Bruising | | | | | | |
| Hematoma | | | | | | |
| Edema | | | | | | |
| Other | | | | | | |

Figure 3-5: Proportion of subjects with observed anticipated injection related reactions (to any intensity level) after first treatment with Sculptra (both sides of the face combined), Safety population

Same tables and figure for treatment sessions two, three and four

Table 3-44: Brief summary of all AEs, Main study, Safety population

| | So | culptra, N=2 | XX | C | ontrol, N=Y | Y |
|---|---|---|---|---|---|---|
| | Subjects<br>n % | | Events<br># | Subjects<br>n % | | Events<br># |
| Adverse Events reported, total | | | | | | |
| Total, serious | | | | | | |
| Total, non-serious | | | | | | |
| AEs related to injection procedure and/or product, total | | | | | | |
| Serious | | | | | | |
| Non-serious | | | | | | |
| Unrelated AEs, total | | | | | | |
| Serious | | | | | | |
| Non-serious | | | | | | |
| Subjects with no AE reported | | | | | | |

 $<sup>\</sup>frac{0}{0} = (n/N)*100$ 

Table 3-45: Related Adverse Events by MedDRA SOC and preferred term,

Main study, subjects randomized to Sculptra, Safety population

| Drimorry SOC | Dun farma d Tarres | Subjects | | Events | Maximal Intensity | | |
|---|---|---|---|---|---|---|---|
| Primary SOC | Preferred Term | n | % | # | Mild | Moderate | Severe |
| Total | | | | | | | |

 $<sup>\</sup>frac{1}{\%}$  = (n/number of subjects in the Safety population)\*100

Print date: 2023-11-27 15:03

GALDERMA

Title
43CHSA1803 Statistical Analysis Plan - Sculptra China

MA-40407

Table 3-46: Related Adverse Events by MedDRA SOC and preferred term, by treatment session, Main study, subjects randomized to Sculptra, Safety population

| Visit | Drim our COC | Preferred Term | Sub | jects | Events | N | Iaximal Intensi | ty |
|---|---|---|---|---|---|---|---|---|
| VISIT | Primary SOC | Preferred Term | n | % | # | Mild | Moderate | Severe |
| Baseline / Treatment 1 | | | | | | | | |
| Treatment 2 (optional) | | | | | | | | |
| Treatment 3 (optional) | | | | | | | | |
| Treatment 4 (optional) | | | | | | | | |

<sup>%</sup> = (n/number of subjects in the Safety population)\*100

Doc id 43CHSA1803 Statistical Analysis Plan - Sculptra China ♣ GALDERMA **MA-40407** 

Print date:

2023-11-27 15:03

Table 3-47: Time to onset from last treatment of related AEs,

| Main study, subjects randomized to | viain study, subjects randomized to Sculptra, Safety population | | | | | |
|---|---|---|---|---|---|---|
| Preferred term | | Time to onset (days) | | | | |
| Treferred term | n | Mean | SD | Min | Median | Max |
| Total | | | | | | |

NA = Not Applicable

Table 3-48: Duration of related AEs,

Main study, subjects randomized to Sculptra, Safety population

| | to Scuiptia, Saicty population | | | | | |
|---|---|---|---|---|---|---|
| Preferred term | Duration (days) | | | | | |
| | n | Mean | SD | Min | Median | Max |
| Total | | | | | | |

NA = Not Applicable

Table 3-49: Action taken of related AEs,

Main study, subjects randomized to Sculptra, Safety population

| riam study, subjects randomized to Scuiptra, Safety population | | | | |
|---|---|---|---|---|
| | Action taken | | | |
| Preferred term | None | Medication<br>treatment | Non-<br>pharmacological<br>treatment or other<br>procedures / tests | Withdrawn |
| Total | | | | |

Table 3-50: Unrelated Adverse Events by MedDRA SOC and preferred term,

Main study, Subjects randomized to Sculptra, Safety population

| Primary SOC Preferred | Preferred Term | Sub | | Events | Maximal Intensity | | |
|---|---|---|---|---|---|---|---|
| Filliary SOC | ary SOC Preferred Term | | % | # | Mild | Moderate | Severe |
| Total | | | | | | | |

<sup>% = (</sup>n/number of subjects in the Safety population)\*100

Table 3-51: Unrelated Adverse Events by MedDRA SOC and preferred term, Main study, Subjects randomized to no-treatment control, Safety population

| Primary SOC | Preferred Term | Subjects | | Events | Maximal Intensity | | |
|---|---|---|---|---|---|---|---|
| | | n | % | # | Mild | Moderate | Severe |
| Total | | | | | | | |

<sup>% = (</sup>n/number of subjects in the Safety population)\*100

# AE tables for Extension phase

Same tables as above when applicable

# AE tables for Combined phases

Same tables as above when applicable

# Group A

The same tables as for Group B, when applicable

Title
43CHSA1803 Statistical Analysis Plan - Sculptra China Doc id ♣ GALDERMA **MA-40407** 

# SIGNATURES PAGE

Print date:

2023-11-27 15:03

| Date | Signed by |
|------------------|------------------------------|
| 2019-10-23 07:15 | |
| Justification | Approved by Owner |
| 2019-10-23 08:02 | |
| Justification | Approved by Technical Expert |
| 2019-10-23 08:29 | PPD |
| Justification | Approved by Technical Expert |
| 2019-10-24 08:59 | |
| Justification | Approved by Technical Expert |